CLINICAL TRIAL: NCT03100578
Title: Randomized Multicenter Study Comparing Plastic Stents and Self-expanding Metallic Stents Used in the Eus-guided Transmural Drainage of Walled-off Pancreatic Necrosis.
Brief Title: EUS-guided Transmural Drainage of Walled-off Pancreatic Necrosis: Plastic vs Metallic Protesis.
Acronym: PROMETHEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Carlos III Health Institute (Other Government); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Principal Investigator, Joan B Gornals, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROMETHEUS
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Pancreas Necrosis; Pancreatic Collection
Keywords: PANCREAS; ENDOSCOPIC INTERVENTION; PLASTIC STENT; SELF EXPANDING METALLIC STENT; ENDOSCOPIC TRANSMURAL DRAINAGE; WALLED OFF PANCREATIC NECROSIS
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLASTIC STENT (Experimental): Endoscopic double pigtail plastic stent, with formal indication on pancreatic collection, according to the instruction forms of the manufacturer.
  Interventions associated:
  EUS-guided transmural drainage of pancretic collection: PLASTIC STENT.
  Interventions: Device: WOPN TRANSMURAL DRAINAGE: PLASTIC STENT
- SELF EXPANDABLE METALLIC STENT (Active Comparator): Lumen apposing metal stent with formal indicaction on pancreatic collection, according to the manufacturer instruction forms.
  Interventions associated:
  EUS-guided transmural drainage of pancretic collection: METALLIC STENT.
  Interventions: Device: WOPN TRANSMURAL DRAINAGE: METALLIC STENT

INTERVENTIONS:
Device: WOPN TRANSMURAL DRAINAGE: PLASTIC STENT — Endoscopic ultrasound-guided transmural drainage of walled-off pancreatic necrosis:
  The pancreatic collection will be located with the linear echoendoscope, and we will proceed to choose an optimal area to perform the puncture guided by EUS; with the absence of intervening vessels.
  This collection will be punctured with a 19 G needle or with an electrocautery device directly. Guidance will be advanced through the needle and the ostomy will proceed according to the routine of the experienced endoscopist.
  Placement of a plastic double pigtail, 5-10 cm in length, diameters 7-8,5-10 Fr. Minimum one 10 Fr prosthesis.
  Arm associated: PLASTIC STENT
  Arms: PLASTIC STENT
Device: WOPN TRANSMURAL DRAINAGE: METALLIC STENT — Endoscopic ultrasound-guided transmural drainage of walled-off pancreatic necrosis:
  The pancreatic collection will be located with the linear echoendoscope, and we will proceed to choose an optimal area to perform the puncture guided by EUS; with the absence of intervening vessels.
  This collection will be punctured with a 19 G needle or with an electrocautery device directly. Guidance will be advanced through the needle and the ostomy will proceed according to the routine of the experienced endoscopist.
  Placement of a metal self-expanding fully covered luminal apposition stent: 10, 15 or 20 mm diameter.
  Arm associated: SELF EXPANDABLE METALLIC STENT
  Arms: SELF EXPANDABLE METALLIC STENT

SUMMARY:
Randomized multicenter study comparing plastic stents and self-expanding metallic stents in the eus-guided transmural drainage of walled-off pancreatic necrosis.

Spanish centers partners of the spanish society of digestive endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Patient with indication (ASGE, Jacobson BC, GIE2005;) of pancreatic collection drainage type WALLED-OFF PANCREATIC NECROSIS * as a local complication of previous acute pancreatitis.
* Patient trained to understand and / or sign informed consent
* Patient who understands the type of study and will comply with all follow-up of complementary tests during its duration

Exclusion Criteria:

* Pregnancy or breastfeeding
* Severe coagulation disorder: INR> 1.5 not correctable with plasma and / or platelet administration <50,000 / mm3
* Asymptomatic patients, with no clinical indication of drainage, except for those with vascular involvement due to compression (eg stenosis, splenic vessels with collateral circulation, and risk of bleeding)
* Non-identification of solid content during the Endoscopic Ultrasound of the procedure
* No informed consent
* In the case of patients with mental retardation, without the ability to understand the nature and possible consequences of the study, except for the existence of a legal representative
* Patients unable to maintain posterior follow-up (lack of adherence)
* Situations that do not allow the practice of a high digestive endoscopy (eg, stenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
RADIOLOGICAL SUCCESS | 4 weeks
  Radiological success at 4 weeks after the interventional procedure: reduction size of the wopn at least 50%.

SECONDARY OUTCOMES:
CLINICAL SUCCESS | 4 month
  Evaluate the long-term clinical success (4 months) (metallic vs. plastic) determined by the total resolution or <3cm of the WOPN, releated with clinical improvement.
TECHNICAL ASPECTS | 1st day
  Evaluate the technical success, duration of the procedure and level of difficulty.
INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS [SAFETY AND TOLERABILITY] | 1st day, 24h, 7 days, 4 weeks, 8 weeks, 4 month, 6 month, 8 month, 12 month
  Assess safety: complications (immediate, early and late)
RECURRENCES | 4 weeks, 8 weeks, 4 month, 6 month, 8 month, 12 month
  Evaluate recurrences
COSTS ANALYSIS | 12 month
  Evaluate the costs between the two types of strategy

OTHER OUTCOMES:
TECHNICAL ASPECTS | 1st day
  Technical success: Correct release of the prosthesis (plastic or metallic) and drainage of the WOPN.
TECHNICAL ASPECTS | 1st day
  Duration of the procedure: Minutes
TECHNICAL ASPECTS | 1st day
  Level of difficulty: Easy, Medium, Hard, Very hard

CONTACTS AND LOCATIONS:
Overall Officials: JOAN B GORNALS, MD, PhD, Principal Investigator — Hospital Universitari de Bellvitge - IDIBELL
Locations (8):
- Spain (8):
  - Hospital Arnau de Vilanova, Lleida, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital San Juan de Dios, Pamplona, Navarre
  - Hospital Universitario Río Hortega, Valladolid, Valldolid
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gornals JB, Velasquez-Rodriguez JG, Bas-Cutrina F, Garcia Garcia De Paredes A, Esteban JM, Teran A, Gonzalez-Huix F, Perez-Miranda M, Guarner-Argente C, Vila JJ, Garcia-Sumalla A, Foruny JR, Fisac-Vazquez J, Moris M, Miquel-Salas I, De-la-Serna Higuera C, Murzi-Pulgar M, Sanchez-Yague A, Salord S, Ruiz-Osuna S, Busquets J, Sanllorente-Melenchon M, Videla S, Moreno R, Tebe-Cordomi C, Hereu P, Vazquez-Sequeiros E; Spanish Working Group on Pancreatic Collection Therapy. Plastic pigtail vs lumen-apposing metal stents for drainage of walled-off necrosis (PROMETHEUS study): an open-label, multicenter randomized trial. Surg Endosc. 2024 Apr;38(4):2148-2159. doi: 10.1007/s00464-024-10699-w. Epub 2024 Mar 6. PMID 38448625
- [Derived] Gornals JB, Perez-Miranda M, Vazquez-Sequeiros E, Vila J, Esteban JM, Gonzalez-Huix F, Guarner-Argente C, Sanchez-Yague A, Teran A, Bas-Cutrina F, De La Serna C, De Paredes AG, Ballester R, Velasquez-Rodriguez J, Salord S, Tebe C, Hereu P, Videla S; Spanish Working Group on Pancreatic Collection Therapy. Multicenter study of plastic vs. self-expanding metal stents in endoscopic ultrasound-guided drainage of walled-off pancreatic necrosis - PROMETHEUS: a randomized controlled trial protocol. Trials. 2019 Dec 30;20(1):791. doi: 10.1186/s13063-019-3988-x. PMID 31888751